CLINICAL TRIAL: NCT07331805
Title: Randomized, Multicenter, Non-inferiority Clinical Trial to Design a Conservative Strategy for the Treatment of Primary Spontaneous Pneumothorax (PSP)
Brief Title: Conservative Management in Primary Spontaneous Pneumothorax: a Multicenter Randomized Non-inferiority Study
Acronym: CONNEP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Carlos Molero-Cano, Residente de Cirugía General y del Aparato Digestivo, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CONNEP_ 2025/3006
Record Dates: First submitted 2025-09-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-11

CONDITIONS: Primary Spontaneous Pneumothorax (PSP); Conservative Management (Active Observation)
Keywords: Primary Spontaneous Pneumothorax (PSP); Conservative management; Active observation / No initial intervention; Chest tube drainage (standard care); Complete lung re-expansion at 8 weeks; Chest X-ray; Collins method (size estimation); Clinical stability (stable PSP); Recurrence (up to 2 years); Quality of life and cost-effectiveness
MeSH Terms: conditions — Pneumothorax; Recurrence | interventions — Conservative Treatment

STUDY DESIGN:
Intervention Model Description: Randomized, parallel-assignment, multicenter, open-label, non-inferiority clinical trial with two arms (conservative management vs. chest tube), primary purpose: treatment.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative management (active observation) (Experimental): After randomization, participants remain under observation with a repeat chest X-ray ≥4 hours after the diagnostic film. If clinical and radiographic stability persists, they are discharged with structured outpatient follow-up: approximately 1-week review with a pre-visit X-ray, then every ~2 weeks until radiographic resolution (up to about 8 weeks of conservative management if not resolved earlier). Rescue chest tube is performed at any time if clinical deterioration or radiographic progression occurs.
  Interventions: Other: Conservative management (active observation)
- Procedure: Chest tube drainage (Active Comparator): After randomization, participants undergo chest tube insertion per usual care with hospital admission. Drain management and removal follow standard clinical criteria. After discharge, participants attend routine outpatient follow-up with chest X-rays to document resolution and to record complications, additional procedures, and length of stay.
  Interventions: Procedure: Chest tube drainage

INTERVENTIONS:
Other: Conservative management (active observation) — Initial in-hospital observation with a repeat chest X-ray ≥4 hours after the diagnostic film. If clinical and radiographic stability persists, discharge home with structured outpatient follow-up (≈1 week, then about every 2 weeks) until radiographic resolution (up to ~8 weeks if not resolved earlier). Rescue chest tube at any time for clinical deterioration or radiographic progression.
  Arms: Conservative management (active observation)
Procedure: Chest tube drainage — Chest tube insertion per usual care with hospital admission. Drain management and removal follow standard clinical criteria. After discharge, routine outpatient follow-up with chest X-rays documents resolution and tracks complications, additional procedures, and length of stay.
  Arms: Procedure: Chest tube drainage

SUMMARY:
The goal of this randomized clinical trial is to find out whether a conservative management strategy (active observation without an initial invasive procedure) can treat as effectively as the standard treatment with chest tube drainage in adults with a large primary spontaneous pneumothorax who are clinically stable. Participants include men and women 18 to 60 years old with a lung collapse ≥30% (by Collins method).

The main questions are:

* Is conservative management not inferior to chest tube drainage for achieving complete lung re-expansion at 8 weeks (on chest X-ray)?
* What are the differences between the two strategies in complications, recurrence at 2 years, quality of life, length of hospital stay, number of additional procedures, and healthcare costs?

Comparison groups:

* Conservative management: in-hospital observation with a control chest X-ray no earlier than 4 hours; if the person remains stable, discharge home with scheduled outpatient follow-up and serial X-rays until resolution.
* Standard treatment (chest tube): chest tube placement and hospital admission; discharge based on clinical progress with routine outpatient follow-up.

Researchers will compare both groups to see whether conservative management works just as well to resolve the pneumothorax at 8 weeks and whether it leads to fewer complications, shorter hospital stays, better quality of life, and lower costs.

What will participants be asked to do? Review the participant information sheet and sign informed consent.

Be randomized by computer (REDCap) to either conservative management or chest tube drainage.

Depending on the assigned group:

* Conservative group: remain under observation initially, have a chest X-ray at ≥4 hours; if still stable, go home with clinic visits (about 1 week after discharge and then every ~2 weeks) until the pneumothorax has resolved.
* Chest tube group: undergo chest tube insertion, stay in the hospital, and attend routine outpatient follow-up after discharge.

Undergo chest X-rays interpreted by the clinical team (with centralized review procedures).

Complete brief symptom assessments, quality-of-life questionnaires (e.g., EQ-5D-5L), and attend follow-up visits or phone calls for up to 2 years to check for recurrences.

This is a multicenter study conducted in several hospitals in Spain. The planned sample size is 436 participants (218 per group), with a non-inferiority margin of 5% and the primary assessment at 8 weeks.

DETAILED DESCRIPTION:
Background and Rationale

Primary spontaneous pneumothorax (PSP) commonly affects young, otherwise healthy individuals. Large PSP has traditionally been managed with chest tube drainage and hospital admission, which can cause pain, longer stays, and procedure-related complications. Emerging evidence and guideline trends suggest that, in clinically stable, minimally symptomatic patients, a conservative strategy (no immediate invasive procedure) may be as effective as invasive options while reducing complications and improving patient experience. However, the current evidence base remains limited, justifying a multicenter randomized trial to rigorously compare both strategies.

This protocol uses the Collins method on chest radiography to estimate pneumothorax size because it correlates with CT-based estimates and is practical for routine care.

Primary Objective

To demonstrate the non-inferiority of conservative management compared with chest tube drainage in achieving complete lung re-expansion at 8 weeks, defined as no pleural air on chest X-ray.

Secondary Objectives

Between strategies, to compare: treatment-related complications (e.g., bleeding, infection, persistent air leak, tension physiology), recurrence up to 2 years, quality of life and patient satisfaction (including EQ-5D-5L), time to clinical and radiographic resolution, length of hospital stay, number of invasive procedures, days of work/disability, drainage characteristics in the invasive arm, healthcare costs, and site-level variation (e.g., hospitals with or without thoracic surgery on site).

Study Design

Prospective, randomized, multicenter, non-inferiority clinical trial comparing no initial intervention (conservative strategy) versus standard treatment (chest tube drainage) in large PSP with clinical stability. The trial assesses effectiveness, safety, quality of life, and cost-effectiveness.

Sponsor and Sites

The study is sponsored by an academic research institute. Multiple sites across Spain are currently recruiting; specific site names are not listed here.

Target Population

Adults with large PSP who are clinically stable and eligible for conservative management within the trial context. (Detailed inclusion/exclusion criteria are provided in the Eligibility section of the registry and are not duplicated here.)

Interventions

Conservative management (experimental):

Initial observation in the hospital with a control chest X-ray ≥4 hours after the diagnostic film.

If clinical and radiographic stability persists, discharge home with scheduled outpatient follow-up: approximately 1-week review with pre-visit chest X-ray, then every ~2 weeks until radiographic resolution (up to 8 weeks of conservative management if no earlier resolution).

Rescue with chest tube if clinical deterioration or radiographic progression occurs at any point.

Standard treatment (comparator):

Chest tube insertion per usual care and hospital admission.

Routine outpatient follow-up after discharge.

Randomization and Blinding

Central randomization is performed via a secure electronic system (e.g., REDCap) with concealed allocation. Given the nature of the interventions (no procedure vs. chest tube), the trial is open-label for participants and clinicians; the protocol specifies standardized follow-up procedures and quality checks to minimize assessment bias.

Outcomes and Assessments

Primary outcome: Complete lung re-expansion at 8 weeks on chest X-ray (no pleural air). Imaging is read by the clinical team with predefined verification procedures to support consistency.

Key secondary outcomes: Complications, recurrence to 2 years, quality of life (including EQ-5D-5L), time to clinical/radiographic resolution, hospital length of stay, number of invasive procedures, days of work/disability, drainage parameters (in the invasive arm), healthcare costs, and exploratory comparisons by site type.

Sample Size and Statistical Plan

Planned enrollment is 436 participants (218 per group), assuming 8-week resolution rates of approximately 98% (drainage) and 97% (conservative), a non-inferiority margin of 5%, α=0.05, and β=0.20. Analyses will follow intention-to-treat and per-protocol principles (for the latter, participants randomized to conservative management who require chest tube due to progression/deterioration at the ≥4-hour assessment are analyzed within the interventional framework as specified). A mid-trial analysis is planned at ~50% enrollment with appropriate statistical safeguards. A health economic evaluation will estimate incremental costs and outcomes between strategies.

Procedures and Follow-up Schedule

Screening and consent at diagnosis (emergency department or inpatient setting).

Randomization via the electronic system and initiation of assigned management.

Conservative arm: observation and ≥4-hour repeat film; if stable, discharge with structured follow-up (≈1 week, then every ~2 weeks) including chest X-rays until resolution or 8 weeks.

Chest tube arm: hospital admission with standard care and routine outpatient follow-up after discharge.

Long-term follow-up for recurrence up to 2 years (clinic visits and/or phone contacts per schedule).

Data Management and Quality Assurance

Participating sites are trained to deliver the protocol consistently. The coordinating center conducts periodic internal audits/monitoring of enrollment, protocol adherence, data completeness, and safety reporting. Data are captured prospectively in a secure electronic database (e.g., REDCap) with role-based access, validation checks, and audit trails.

Network Size and Timelines

A national network is active. Assuming an average of ~1.5-2 participants per site per month and ~12 active sites, anticipated accrual is ~18-24 participants/month, yielding a ~20-24-month recruitment period (with allowances for start-up variability). Total on-study time includes follow-up for the primary endpoint at 8 weeks and recurrence monitoring to 2 years.

Ethics and Safety

Both strategies are accepted standards of care for stable PSP; the study does not introduce experimental procedures. Participant confidentiality follows applicable regulations (e.g., GDPR). Consent forms and linkage files are stored securely; access is limited to authorized study personnel, auditors, and regulators as required. Safety oversight includes predefined criteria for rescue intervention and adverse event reporting.

Clinical Relevance

If non-inferiority of conservative management is confirmed, the results could reduce invasive procedures and hospital stays, improve patient-reported outcomes, and optimize resource use in PSP-while maintaining comparable resolution rates and safety. Findings would support more selective use of chest tubes, align practice with up-to-date evidence, and incorporate patient preferences when clinically appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Age: >18 and ≤60 years at the time of enrollment.
* Diagnosis: Primary spontaneous pneumothorax of large size (lung collapse ≥30% by the Collins method on chest X-ray).
* Episode type: Any episode of primary spontaneous pneumothorax.
* Clinical stability suitable for observation without immediate intervention: Systolic BP >90 mmHg, heart rate <140 bpm, oxygen saturation >90% (with supplemental oxygen if needed), respiratory rate 15-30 breaths/min.
* Consent: Has read and understood the participant information sheet and signed informed consent.

Exclusion Criteria:

* Pre-existing lung disease that may predispose to pneumothorax (e.g., COPD, cystic fibrosis, interstitial lung disease, tuberculosis, pulmonary neoplasm).
* Indication for urgent thoracic surgery (e.g., imaging highly suggestive of giant bullae/blebs requiring immediate surgical intervention).
* Pregnancy or breastfeeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 436 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Complete lung re-expansion on chest X-ray | 8 weeks after randomization.
  Proportion of participants with no pleural air on the 8-week chest X-ray (definition of complete radiographic resolution).

SECONDARY OUTCOMES:
Treatment-related complications | Procedure- or management-related adverse events (e.g., bleeding, infection, persistent air leak, need for reintervention or surgery), prospectively recorded.
  Up to 24 weeks
Recurrence of pneumothorax. | Up to 2 years after resolution of the index episode.
  New ipsilateral pneumothorax occurring after documented complete resolution of the index event.
Health-Related Quality of Life Assessed by EQ-5D-5L | Up to 24 weeks
  Changes in health-related quality of life measured using the EuroQol EQ-5D-5L questionnaire. Scores range from -0.281 to 1.000, with higher scores indicating better quality of life. Comparison between conservative management and chest tube drainage.

IPD SHARING:
Plan to Share IPD: No